CLINICAL TRIAL: NCT01341379
Title: Increasing Ureagenesis in Inborn Errors of Metabolism With N-Carbamylglutamate
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Marc Yudkoff, Division Chief, Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-007806; R01HD058567 (NIH)
Record Dates: First submitted 2011-04-22; First posted 2011-04-25 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Urea Cycle Disorders, Inborn; Inborn Errors of Metabolism; Propionic Acidemia; Methylmalonic Acidemia; Carbamyl Phosphate Synthetase Deficiency
Keywords: Ureagenesis; Urea cycle; Inborn errors of metabolism
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Metabolism, Inborn Errors; Propionic Acidemia; Methylmalonic acidemia; Carbamoyl-Phosphate Synthase I Deficiency Disease | interventions — N-carbamylglutamate; carglumic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- N-carbamylglutamate (Carbaglu) (Experimental)
  Interventions: Drug: N-carbamylglutamate

INTERVENTIONS:
Drug: N-carbamylglutamate — N-carbamylglutamate: 200 mg/kg/day for 3 days, divided into 4 daily oral doses
  Other Names: Carbaglu

SUMMARY:
Hyperammonemia, which can cause brain damage, occurs in many different kinds of inborn errors of metabolism. The investigators propose to determine if short-term (3 day) treatment with N-carbamylglutamate can diminish hyperammonemia by enhancing ureagenesis in these patients. The investigators propose here a short-term (3 day) trial. If it succeeds, the investigators would consider more extensive long-term studies of the drug.

DETAILED DESCRIPTION:
* To determine whether brief (3 day) treatment with N-carbamylglutamate can improve ureagenesis in adult healthy controls and patients with the following inborn errors of metabolism: N-acetylglutamate synthetase deficiency, propionic acidemia, methylmalonic acidemia, carbamylphosphate synthase deficiency, ornithine transcarbamylase deficiency and the syndrome of hyperammonemia, hypoglycemia and hyperinsulinemia (HHH Syndrome).
* To determine if such treatment improves other indicators of abnormal nitrogen metabolism such as elevated blood levels of glutamine, glycine and alanine.

ELIGIBILITY:
Inclusion Criteria:

* Age range: males or females, ages 3 years - 70 years
* Condition(s): N-acetylglutamate synthetase deficiency, propionic acidemia, methylmalonic acidemia, carbamylphosphate synthase deficiency, ornithine transcarbamylase deficiency and the syndrome of hyperammonemia, hypoglycemia and hyperinsulinemia.
* In addition, healthy volunteers will be studied (ages 18 years - 50 years).

Exclusion Criteria:

* Acutely ill on day of study (fever, evidence of hyperammonemia - ataxia, worsening obtundation, focal neurologic signs, seizures, increased intracranial pressure, vomiting, signs of acute respiratory or enteric illness, headache, confusion, disorientation, acute personality change).
* Girls 11 years of age must have a negative urine/serum pregnancy test within 1 week prior to testing unless having a menstrual period during week of test
* Lactating females
* Hyperammonemia probably refractory to N-carbamylglutamate: other urea cycle disorders (UCD), lysinuric protein intolerance, mitochondrial disorders, congenital lactic acidemia, fatty acid oxidation defects or primary liver disease.
* Amount of blood necessary for study exceeds safe limits.
* Any investigational drug use within 30 days prior to enrollment.
* Parents/guardians or subjects who, in the opinion of the PI, may be non-compliant with study schedules or procedures.
* Subjects who do not meet all the enrollment criteria may not be enrolled. Any violations of these criteria will be reported in accordance with Institutional Review Board (IRB) Policies and Procedures.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Rate of ureagenesis | 3 days
  Goal is to determine whether a 3 day trial of N-carbamylglutamate increases ureagenesis in patients with urea cycle defects and other inborn errors of metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Yudkoff, MD, Principal Investigator — Children's Hospital of Philadelphia

REFERENCES:
- [Result] Ah Mew N, McCarter R, Daikhin Y, Nissim I, Yudkoff M, Tuchman M. N-carbamylglutamate augments ureagenesis and reduces ammonia and glutamine in propionic acidemia. Pediatrics. 2010 Jul;126(1):e208-14. doi: 10.1542/peds.2010-0008. Epub 2010 Jun 21. PMID 20566609
- [Result] Yudkoff M, Ah Mew N, Daikhin Y, Horyn O, Nissim I, Nissim I, Payan I, Tuchman M. Measuring in vivo ureagenesis with stable isotopes. Mol Genet Metab. 2010;100 Suppl 1(Suppl 1):S37-41. doi: 10.1016/j.ymgme.2010.02.017. Epub 2010 Feb 26. PMID 20338795
- [Result] Ah Mew N, Payan I, Daikhin Y, Nissim I, Nissim I, Tuchman M, Yudkoff M. Effects of a single dose of N-carbamylglutamate on the rate of ureagenesis. Mol Genet Metab. 2009 Dec;98(4):325-30. doi: 10.1016/j.ymgme.2009.07.010. Epub 2009 Jul 14. PMID 19660971
- [Result] Tuchman M, Caldovic L, Daikhin Y, Horyn O, Nissim I, Nissim I, Korson M, Burton B, Yudkoff M. N-carbamylglutamate markedly enhances ureagenesis in N-acetylglutamate deficiency and propionic acidemia as measured by isotopic incorporation and blood biomarkers. Pediatr Res. 2008 Aug;64(2):213-7. doi: 10.1203/PDR.0b013e318179454b. PMID 18414145